CLINICAL TRIAL: NCT07318415
Title: Quantitative Assessment of Vaginal Tissue Response to Intravaginal Brachytherapy With Multiparametric Ultrasound Imaging (mpUS)
Brief Title: A Study of Multiparametric Ultrasound Imaging (mpUS) for People With Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-157
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: stage I-II endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Masking Description: This will be a prospective, single center clinical study with 10 patients with endometrial cancer to test the feasibility of using mpUS to characterize the vaginal tissue response to IVRT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiparametric Ultrasound Imaging (mpUS) (Experimental): All participants in this study will receive standard intravaginal brachytherapy (IVRT) and multiparametric ultrasound (mpUS) imaging right before IVRT, right after the last IVRT, and at 3, 6 and 12 months after IVRT.
  Interventions: Diagnostic Test: Multiparametric Ultrasound Imaging; Other: The vaginal assessment score (VAS)

INTERVENTIONS:
Diagnostic Test: Multiparametric Ultrasound Imaging — multiparametric ultrasound (mpUS) imaging right before IVRT, right after the last IVRT, and at 3, 6 and 12 months after IVRT
Other: The vaginal assessment score (VAS) — The vaginal assessment score (VAS) is a four-item measure that is administered to the patient to quantify and rate (none, mild, moderate, or severe) their perception of dryness, soreness, irritation, and pain (dyspareunia or painfulness to touch with external stimulation).

SUMMARY:
The researchers are doing this study to see how well multiparametric ultrasound (mpUS) imaging can evaluate vaginal tissue before and after IVRT. IVRT is routinely used to treat endometrial cancer but can cause damage to the vaginal tissue (vaginal toxicity). Side effects of vaginal toxicity can include vaginal dryness, itching, soreness, discharge, narrowing or shortening of the vagina (stenosis), and vaginal fibrosis (hardening), which can affect sexual function. The researchers will also look at whether participants are able to complete (tolerate) all mpUS imaging for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with a primary endometrial carcinoma. The following histologic subtypes are eligible for inclusion: endometrioid, serious, clear cell, dedifferentiated/undifferentiated, mixed epithelial, adenocarcinoma not otherwise specified, and carcinosarcoma
* Initial surgical treatment must have included hysterectomy, bilateral salpingo-oophorectomy, and pelvic lymph node assessment with either sentinel lymph node mapping/sampling or pelvic lymph node dissection. Surgical assessment of the para-aortic lymph nodes is not required
* Patients must have had a complete surgical resection with negative margins and no residual gross disease after surgery
* Patients must have FIGO (2009) stage I-II disease (per surgical staging)
* Age ≥ 18 years
* Patients must be able to start radiotherapy within 12 weeks from date of surgery

Exclusion Criteria:

* Patients receiving chemotherapy or hormonal therapy
* A prior or concurrent malignancy whose natural history or treatment would interfere with the toxicity or efficacy assessment of IVRT
* Prior pelvic radiotherapy
* Active genitourinary infection requiring antibiotics, except for uncomplicated urinary tract infection
* History of active inflammatory bowel disease requiring treatment, including Crohn's disease and ulcerative colitis
* Concurrent psychiatric or medical condition or disease which, per investigator judgement, would make them unsuitable candidates for study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer
Enrollment: 10 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
feasibility of B-mode ultrasound imaging | 1 year
  B-mode feasibility is defined as the ability to visualize/quantify vaginal wall thickness and echogenicity at baseline and immediately following the last IVRT treatment in 6 out of 10 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kaled Alektiar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org